CLINICAL TRIAL: NCT06055504
Title: Study of Personalized Allocation of Defibrillators in Non-ischemic Heart Failure (SPANISH-1)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPANISH-1
Record Dates: First submitted 2023-04-24; First posted 2023-09-26 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Non-ischemic Dilated Cardiomyopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Strategy (Other)
  Interventions: Other: Control Strategy
- Personalized precision ICD implantation Strategy based in genetic findings and CMR results (Experimental)
  Interventions: Other: Personalized precision ICD implantation Strategy based in genetic findings and CMR results

INTERVENTIONS:
Other: Control Strategy — ICDs will be implanted in all patients according to current recommendations
  Arms: Control Strategy
Other: Personalized precision ICD implantation Strategy based in genetic findings and CMR results — Patients allocated to the intervention strategy will receive an ICD according to genetic and CMR results. ICD implantation criteria in patients allocated to the personalised strategy group will be the presence of either a DCM-causing pathogenic or likely pathogenic genetic variants or LGE in CMR. Patients without DCM-associated genetic variants and without LGE on CMR will not receive standard treatment but an ICD will not be implanted on them.
  Arms: Personalized precision ICD implantation Strategy based in genetic findings and CMR results

SUMMARY:
Prospective, randomised, multicentre, open-label study to assess the non-inferiority of a personalised precision strategy for Sudden Cardiac Death (SCD) prevention in patients with non-ischemic dilated cardiomyopathy with Left Ventricular Ejection Fraction (LVEF) ≤35%

DETAILED DESCRIPTION:
Prospective, randomised, multicentre, open-label study to assess the non-inferiority of a personalised precision strategy for SCD prevention in patients with non-ischemic dilated cardiomyopathy with LVEF≤35%

Randomization will be 1:1 and patients are allocated to either control strategy or intervention strategy.

In the control strategy group, patients will get an Implantable Cardioverter Defibrillator (ICD) implanted. Patients allocated to the intervention strategy will receive an ICD according to genetic and CMR results. ICD implantation criteria in patients allocated to the personalised strategy group will be the presence of either a Dilated Cardiomyopathy DCM-causing pathogenic or likely pathogenic genetic variants or Late Gadolinium Enhancement (LGE) in Cardiac Magnetic Resonance (CMR). Patients without DCM-associated genetic variants and without LGE on CMR will not receive standard treatment but an ICD will not be implanted on them.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of screening.
* Previously established diagnosis of Non-ischemic DCM
* Optimised medical treatment at maximum tolerated doses for at least 3 months prior to the screening date.
* NYHA functional class II-III.
* LVEF ≤ 35% documented by CMR as study procedure.
* Life expectancy greater than 12 months.

Exclusion Criteria:

* History of coronary artery disease justifying the presence of ventricular dysfunction, defined as: history of coronary revascularisation or presence of significant coronary stenosis (≥50% in left main or ≥70% in a major epicardial artery) on invasive or non-invasive coronary angiography (coronary CT)
* Left ventricular dysfunction attributed to congenital heart disease, valvular disease, alcohol abuse or chemotherapy.
* Hypertrophic or infiltrative cardiomyopathy, active myocarditis or constrictive pericarditis.
* History of recovered sudden death or sustained ventricular tachycardia.
* NYHA functional class IV.
* Waiting list for cardiac transplantation in emergency 0.
* Receiver of a solid organ transplant (lung, liver, heart or kidney).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Composite end-point of all cause death, hospitalization due to device-related complications, and non-fatal major arrhythmic events. | 4 years

SECONDARY OUTCOMES:
All-cause death | 4 years
SCD | 4 years
Hospitalisation for device-related complications | 4 years
Non-fatal major arrhythmic events | 4 years
cost-effectiveness | 4 years
  Incremental Cost-effectiveness ratio (ICER) of personalized ICD allocation strategy in non-ischemic DCM [ Time Frame: The time horizon of the evaluation will be limited to 4 years ]
  The ICER of the personalized ICD allocation strategy compared with standard strategy is defined as the ratio between the variation in costs and the variation in effectiveness between both strategy groups. In the personalized strategy group, costs will include those related to personalization tests (CMR and genetic analysis) plus costs related to implanting and carrying an ICD (in the number of patients who eventually receive a device). In the control group, costs will include only the latter concept. Costs will be measured in Euros. The variation in effectiveness will be measured both in terms of life years gained, measured in years, and in terms of quality of life gained, measured in QALY. In the first case, ICER will be measured as Euros/year; in the second, it will be measured as Euros/QALY.
Quality of life assessed by KCCQ, EQ-5D and HADS | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Pablo García Pavía, Principal Investigator — H.U. Puerta de Hierro, Majadahonda; Antoni Bayés Genís, Principal Investigator — H.U. Germans Trias i Pujol; Javier Bermejo Thomas, Principal Investigator — H.G.U. Gregorio Marañón; Javier Díez Martínez, Principal Investigator — University of Navarra
Locations (31):
- Spain (31):
  - H.C.U de Santiago de Compostela, Santiago de Compostela, A Coruña
  - H.U. de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Parc Taulí, Sabadell, Barcelona
  - H.U. A Coruña, A Coruña, La Coruña
  - H.U. Puerta de Hierro, Majadahonda, Madrid
  - H.U. Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General Universitario Dr Balmis, Alicante
  - H.U. de la Santa Creu i Sant Pau, Barcelona
  - H. Clinic de Barcelona, Barcelona
  - H.U. Germans Trias i Pujol, Barcelona
  - H.U. Vall d'Hebron, Barcelona
  - H.U. Josep Trueta, Girona
  - H.U. Virgen de las Nieves, Granada
  - Hospital Arnau de Vilanova, Lleida
  - H.G.U. Gregorio Marañón, Madrid
  - H.U. Ramón y Cajal, Madrid
  - H. Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - H.U. 12 de Octubre, Madrid
  - H.U. Virgen de la Victoria, Málaga
  - H.C.U. Virgen de la Arrixaca, Murcia
  - H.U. Son Llátzer, Palma de Mallorca
  - Complejo Hospitalario de Navarra, Pamplona
  - H.U de Salamanca, Salamanca
  - H.U. Virgen del Rocio, Seville
  - Complejo Hospitalario Universitario de Toledo, Toledo
  - H.C.U de Valencia, Valencia
  - H.U. Politécnico de la Fe, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - H.C.U de Valladolid, Valladolid
  - H.U. Miguel Servet, Zaragoza